CLINICAL TRIAL: NCT04512469
Title: A Randomized Controlled Trial Examining the Efficacy of Prophylactic on Lay Mesh Versus Standardized Fascial Closure on Ventral Incisional Hernia Rates in Liver Transplant Patients
Brief Title: Study on the Efficacy of Prophylactic on Lay Mesh in Preventing Post-operative Hernia in Liver Transplant Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Hernia Mesh Liver Transplant
Record Dates: First submitted 2020-07-07; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2019-12

CONDITIONS: Incisional Hernia of Anterior Abdominal Wall
Keywords: liver transplant; incisional hernia
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Intervention Model Description: The research coordinators will identify patients diagnosed with end-stage liver disease who are candidates for liver transplantation for study eligibility (see inclusion and exclusion criteria). Participants will be randomly selected to be included in one of two groups: the control or treatment group. The control group will undergo standard running fascial closure with PDS while the treatment group will undergo this closure plus a low molecular weight mesh extending 3 cm from the fascial incision.
  There will be no alteration to this standard of care schedule for this clinical trial. Data will be collected at every 12-month intervals to rule out clinical evidence of a hernia. The presence of a hernia will be assessed via clinical examination and abdominal ultrasound imaging. If findings from the abdominal ultrasound are inconclusive, a non-contrast CT scan will be performed. The study will end when either the primary or secondary outcomes are reached.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Group (No Intervention): The control group will undergo standard running fascial closure with PDS .
- Treatment Group - Mesh (Experimental): The treatment group will undergo standard running fascial closure with PDS plus a low molecular weight mesh extending 3 cm from the fascial incision.
  Interventions: Device: Low molecular weight mesh

INTERVENTIONS:
Device: Low molecular weight mesh — Following liver implantation, the subcostal incision will be closed using a running fascial closure with absorbable 1-0 Polydioxanone (PDS) suture and staples, with the treatment group also receiving a mesh.
  Arms: Treatment Group - Mesh

SUMMARY:
Study Design: Single-blinded, randomized, prospective clinical trial. Study Population: End-stage liver disease patients' candidates for liver transplantation.

Study procedures: Consenting patients will be divided into two matched groups:

1. CONTROL group - receiving a standard running fascial closure with PDS suture
2. TREATMENT group - receiving a standard running fascial closure with PDS suture PLUS a low molecular weight mesh. The mesh will be secured to the fascia extending 3 cm from the incisional site.

There will be no modifications to routine post-operative wound care in both groups. However, the treatment group will have an additional drain placed at the incision site compared to the control group to reduce the risk of a seroma from placement of the mesh. Wound dressing will be removed on post-op day 2 and the wound will be assessed. Re-application of the dressing will occur thereafter until proper healing of the incision.

An abdominal ultrasound will be done on all study participants at the 1- and 2-year mark postoperatively to look for objective evidence of a ventral incisional hernia. A CT scan will be performed if the abdominal ultrasound findings are inconclusive.

DETAILED DESCRIPTION:
An incisional hernia is a common complication of abdominal surgery with an incidence of 4-20%. Liver transplant patients represent a unique cohort of surgical patients with immediate immune suppression post-operatively. It is presumed that this immune suppression accompanied by significant co-morbidities have led to high incisional ventral hernia rates between 4.9%-34.3%.

A recent 2018 retrospective review of 1044 liver transplant patients identified age >55, high BMI > 25, and immediate rejection were significant risk factors contributing to herniation. However, previously concerning considerations including gender, diagnosis, diabetes, Child-Pugh score, MELD score, donor type, hepato-renal syndrome, varix bleeding, ascites, hepatic encephalopathy, ventilator use, spontaneous bacterial peritonitis (SBP), or bile leak were not identified as significant risk factors. Moreover, the mortality for chronic liver disease patients for elective hernia repair is 3.7% at 90 days and morbidity is 27%. Emergent hernia repair led to 10% 90-day mortality with 60% morbidity. The high incidence of herniation represents a common problem with significant morbidity and mortality post liver transplantation thereby requiring investigating a new preventative solution.

A recent retrospective trial in the colorectal literature identified an institutional incidence of incisional hernia for colorectal patients of 39.9%. They recognized two high-risk populations, obese, and non-obese with a combination of several secondary risk factors. A follow-up prospective cohort study separated all colorectal patients undergoing laparotomy to standardized running PDS closure versus those with BMI>29 (the median in the prior study) and those BMI <29 with >=2 risk factors to include standard closure with an on-lay Ultrapro partially absorb-able mesh covering 3 cm adjacent to the incision placed with double down facial staples followed by a subcutaneous drain. The reported risk factors included BMI, smoking, serum creatinine, hemoglobin, serum albumin, COPD diabetes, immune suppression with steroids or radiation/chemotherapy, and previous midline laparotomy. The results revealed a decrease in the incisional hernia rate from 43.9% to 10% (P=0.0001). This study also concluded the treatment was cost effective and safe.

ELIGIBILITY:
Inclusion Criteria:

• All patients above 18 years of age undergoing liver transplantation

Exclusion Criteria:

* Non consenting patients
* patients with skin or deep tissue infections at the time of surgery
* prior mesh infection from hernia repair will be excluded
* entry into the gastro-intestinal system (i.e., need for hepaticojejunostomy for transplantation versus just a standard biliary-biliary anastomosis)
* prior biliary stent (causes colonization of the biliary track and increases surgical site infection)
* patients that are unstable, requiring pressors, or required >4 units of packed red blood cell transfusions intra-operatively will be excluded as to not prolong surgical time.
* Pregnant women
* Prior incisional hernia/history of IH and repair
* Death within 1-year
* Insufficient follow up
* Connective tissue disorders
* Prior significant wound dehiscence or infection
* Spontaneous bacterial peritonitis
* Primary sclerosing cholangitis (requires roux en y reconstruction thereby entry into the Alimentary track)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Rate of incisional hernia post-operatively | 1 year
  The primary outcome will be incisional hernia rate at 1 year post-operatively.

SECONDARY OUTCOMES:
Rate of incisional hernia post-operatively | 2 years
  Incisional hernia rates at post-operative year 2
Rate of surgical complications | 2 years
  Assess rate of surgical complications as per Clavien Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Anton Skaro, MD, Principal Investigator — Associate Professor - Surgery, Schulich School of Medicine & Dentistry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Argudo N, Pera M, Lopez-Cano M, Hernandez L, Sancho JJ, Grande L, Pereira JA. Selective Mesh Augmentation to Prevent Incisional Hernias in Open Colorectal Surgery Is Safe and Cost-Effective. Front Surg. 2018 Feb 16;5:8. doi: 10.3389/fsurg.2018.00008. eCollection 2018. No abstract available. PMID 29503821
- [Result] Bachir NM, Larson AM. Adult liver transplantation in the United States. Am J Med Sci. 2012 Jun;343(6):462-9. doi: 10.1097/MAJ.0b013e3182308b66. PMID 22683615
- [Result] Bucknall TE, Cox PJ, Ellis H. Burst abdomen and incisional hernia: a prospective study of 1129 major laparotomies. Br Med J (Clin Res Ed). 1982 Mar 27;284(6320):931-3. doi: 10.1136/bmj.284.6320.931. PMID 6279229
- [Result] Israelsson LA, Jonsson T. Incisional hernia after midline laparotomy: a prospective study. Eur J Surg. 1996 Feb;162(2):125-9. PMID 8639725
- [Result] Mudge M, Hughes LE. Incisional hernia: a 10 year prospective study of incidence and attitudes. Br J Surg. 1985 Jan;72(1):70-1. doi: 10.1002/bjs.1800720127. PMID 3155634
- [Result] Pereira JA, Pera M, Grande L. [Incidence of incisional hernia after open and laparoscopic colorectal cancer resection]. Cir Esp. 2013 Jan;91(1):44-9. doi: 10.1016/j.ciresp.2012.05.004. Epub 2012 Jul 4. Spanish. PMID 22769029
- [Result] Piazzese E, Montalti R, Beltempo P, Bertelli R, Puviani L, Pacile V, Nardo B, Cavallari A. Incidence, predisposing factors, and results of surgical treatment of incisional hernia after orthotopic liver transplantation. Transplant Proc. 2004 Dec;36(10):3097-8. doi: 10.1016/j.transproceed.2004.10.047. PMID 15686704
- [Result] Vardanian AJ, Farmer DG, Ghobrial RM, Busuttil RW, Hiatt JR. Incisional hernia after liver transplantation. J Am Coll Surg. 2006 Oct;203(4):421-5. doi: 10.1016/j.jamcollsurg.2006.06.017. Epub 2006 Aug 17. PMID 17000384